CLINICAL TRIAL: NCT01692756
Title: Early Anti-inflammatory Treatment in Patients With Acute ACL Tear
Brief Title: Early Treatment for Acute ACL Tear
Acronym: AAA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cale Jacobs (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor-Investigator, Cale Jacobs, Sponsor/Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-0706
Record Dates: First submitted 2012-09-11; First posted 2012-09-25 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Anterior Cruciate Ligament (ACL) Tears
MeSH Terms: conditions — Lacerations | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Kenalog or Placebo (Experimental): Kenalog® (40mg) or saline placebo injection 1-2 days after ACL injury and 12-14 days later.
  Interventions: Drug: Kenalog or placebo
- Kenalog then placebo (Experimental): Subjects will initially receive 40mg injection of Kenalog® 1-2 days after injury and saline placebo at 12-14 days post injury.
  Interventions: Drug: Kenalog then Placebo
- Kenalog only (Experimental): Subjects will receive two consecutive (40 mg) intra-articular injections of Kenalog®
  Interventions: Drug: Kenalog
- Placebo (Placebo Comparator): subjects will receive two consecutive intra-articular saline placebo injections at the same time periods.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Kenalog or placebo
  Other Names: Drug: Kenalog; Other Names:; triamcinolone acetonide injectable suspension; Drug Placebo (for Kenalog); physiologic Saline solution
  Arms: Kenalog or Placebo
Drug: Kenalog then Placebo
  Other Names: Drug: Kenalog; Other Names:; triamcinolone acetonide injectable suspension; Drug Placebo (for Kenalog); physiologic saline solution
  Arms: Kenalog then placebo
Drug: Kenalog
  Other Names: Drug: Kenalog; Other Names:; triamcinolone acetonide injectable suspension
  Arms: Kenalog only
Drug: Placebo
  Other Names: Drug Placebo (for Kenalog); physiologic saline solution
  Arms: Placebo

SUMMARY:
This research study is the first of its kind and will allow health care professionals and researchers to answer many questions about the reasons why anterior cruciate ligament (ACL) injury leads to knee pain and disability and osteoarthritis. We also hope that this study will be the beginning of new, more powerful and safer drugs to help patients with ACL injuries heal sooner and return to sports or daily activities pain free. Study participants will be recruited from the University of Kentucky and Vanderbilt University.

The purpose of this research is to gather information on how safe and effective Kenalog® is in alleviating knee pain following ACL rupture.

DETAILED DESCRIPTION:
Injury to the knee during sports participation often involves partial of full detachment of the ACL. ACL tears cause pain, swelling and inflammation. While the swelling and inflammation usually goes away in time, individuals with ACL injuries may experience pain and notice knee instability (knee slipping, etc.). Often surgery can repair or replace the ACL within the joint, allowing individuals the ability to walk or run again pain free or participate in sports. Unfortunately, osteoarthritis of the knee, which also causes pain and swelling, can occur in that same knee 10-20 years later for reasons which are not well understood.

In this research study, we hope to prevent and reduce the initial post-operative pain. The reduction of pain will allow for earlier movement of the knee joint and preparation for surgery. It may also reduce the risk to develop osteoarthritis in individuals with ACL injuries by treating them within 1-2 days after their injury.

ELIGIBILITY:
Inclusion Criteria:

* currently participating in sporting activities
* Normal contralateral knee status
* Anterior Cruciate Ligament (ACL) injury occurred while playing a sporting activity

Exclusion Criteria:

* underlying inflammatory disease (i.e. Rheumatoid Arthritis, Psoriatic Arthritis, etc.)
* have been diagnosed with hepatitis B or tuberculosis
* currently have an infection, including infection of the skin
* have a disease that weakens your immune system such as diabetes, cancer, HIV or AIDs
* other major medical condition requiring treatment with immunosuppressant or modulating drugs.
* A history of chronic use of non-steroidal anti-inflammatory drugs
* previous exposure or allergic reaction to Kenalog
* prior knee surgery (Ipsilateral or contralateral)
* have received any investigational drug with 4 weeks of study Visit 1

Ages: 14 Years to 33 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 49 (Actual)
Dates: Start 2013-03; Primary Completion 2017-02-05 (Actual); Study Completion 2017-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Lattermann, MD, Principal Investigator — University of Kentucky, Department of Orthopaedic Surgery
Locations (1):
- UK HeathCare Sports Medicine, Lexington, Kentucky, United States

REFERENCES:
- [Result] Lattermann C, Jacobs CA, Proffitt Bunnell M, Huston LJ, Gammon LG, Johnson DL, Reinke EK, Huebner JL, Kraus VB, Spindler KP. A Multicenter Study of Early Anti-inflammatory Treatment in Patients With Acute Anterior Cruciate Ligament Tear. Am J Sports Med. 2017 Feb;45(2):325-333. doi: 10.1177/0363546516666818. Epub 2016 Oct 7. PMID 28146402
- [Result] Lattermann C, Jacobs CA, Bunnell MP, Jochimsen KN, Abt JP, Reinke EK, Gammon LG, Huebner JL, Kraus VB, Spindler KP. Logistical challenges and design considerations for studies using acute anterior cruciate ligament injury as a potential model for early posttraumatic osteoarthritis. J Orthop Res. 2017 Mar;35(3):641-650. doi: 10.1002/jor.23329. Epub 2016 Jun 30. PMID 27279368
- [Derived] King JD, Rowland G, Villasante Tezanos AG, Warwick J, Kraus VB, Lattermann C, Jacobs CA. Joint Fluid Proteome after Anterior Cruciate Ligament Rupture Reflects an Acute Posttraumatic Inflammatory and Chondrodegenerative State. Cartilage. 2020 Jul;11(3):329-337. doi: 10.1177/1947603518790009. Epub 2018 Jul 22. PMID 30033738

RESULTS

PARTICIPANT FLOW:
Groups:
- Kenalog or Placebo: Kenalog® (40mg) or saline placebo injection 1-2 days after ACL injury and 12-14 days later.
  Kenalog or placebo
- Kenalog Then Placebo: Subjects will initially receive 40mg injection of Kenalog® 1-2 days after injury and saline placebo at 12-14 days post injury.
  Kenalog then Placebo
- Kenalog Only: Subjects will receive two consecutive (40 mg) intra-articular injections of Kenalog®
  Kenalog
- Placebo: subjects will receive two consecutive intra-articular saline placebo injections at the same time periods.
  Placebo
Period: Overall Study
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Started | 12 | 12 | 13 | 12
Completed | 11 | 11 | 11 | 12
Not Completed | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: One patient was lost to follow-up (Group 1). Two patients withdrew prior to receiving treatment (Group 2, Group 3). One patient did not attend first study visit and did not receive allocated intervention (Group 3).
Groups:
- Total: Total of all reporting groups
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo | Total
Number analyzed (Participants) | 11 | 11 | 11 | 12 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.45 (2.99) | 19.60 (4.12) | 24.06 (6.57) | 17.80 (2.14) | 19.9 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 5 | 7 | 19
  Male | 8 | 7 | 6 | 5 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 4 | 6
  White | 10 | 10 | 10 | 8 | 38
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 11 | 12 | 45
Knee Injury and Osteoarthritis Scale (KOOS) Pain Subscale [Mean (Standard Deviation); unit: units on a scale] — KOOS consists of 5 subscales with five questions per scale; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life QOL. The last week is taken into consideration when answering the questions. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The baseline KOOS Pain scores are presented here.
  units on a scale | 49.75 (19.10) | 58.33 (15.42) | 50.25 (24.61) | 46.30 (25.02) | 51.05 (21.2)

OUTCOME MEASURES:

1. Primary Outcome: Participant Pain Assessment
Description: Participants with be given a Visual Analog Scale (VAS) pain assessment questionnaire which scores the participant's perceived pain on a scale of 0-10 were zero is no pain and 10 is the worst pain imaginable. The scale will be administered during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: A total of 4 patients (Group 1 n:1, Group 2 n:1, Group 4 n:2) overlooked completing the VAS. This was not realized until the patients had left the study visit preventing the investigator from collecting the information.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 10 | 10 | 11 | 10
units on a scale | -3.9 (2.8) | -2.2 (2.2) | -3.6 (3.0) | -4.3 (3.2)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = 0.33, Kruskal-Wallis

2. Secondary Outcome: Efficacy of Kenalog to Alleviate Knee Pain
Description: The efficacy of Kenalog with be determined using the Knee Injury and Osteoarthritis Outcome Score (KOOS) instrument. Participants will self-report knee pain and function through the KOOS questionnaire during the initial orthopedic consult and during the pre-op assessment prior to surgery, between 1 and 7 days later. The scale scores range from 100 (no symptoms) to zero (extreme symptoms).
Time Frame: Up to seven days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 11 | 11 | 11 | 12
units on a scale | 37.37 (17.50) | 18.94 (11.02) | 30.56 (23.17) | 28.93 (22.36)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = 0.08, Kruskal-Wallis

3. Secondary Outcome: Synovial Interleukin-1α (IL-1α) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure IL-1α concentration using an immunoassay. Data will be presented as the change in IL-1α concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: The values for 3 patients (Gp1 n:1, Gp 2 n:1, Gp 3 n:1) were below the limits of detection and were not included in the analysis.Two other patients had dry knee aspirations, where the aspiration was performed but no fluid was collected, (Gp 1 n:1, Gp 2 n:1) and 1 patient declined 1 aspiration (Gp 3 n:1) preventing analysis on these patients.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 9 | 9 | 9 | 12
pg/mL | 4.30 (6.59) | 7.68 (13.15) | 1.77 (4.43) | 3.11 (5.03)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = 0.93, Kruskal-Wallis

4. Secondary Outcome: Synovial Interleukin-1β (IL-1β) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure IL-1β concentration using an immunoassay. Data will be presented as the change in IL-1β concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: The values for two patients (Gp1 n:1, Gp 2 n:1) were below the limits of detection and were not included in the analysis. Two other patients had dry knee aspirations, where the aspiration was performed but no fluid was collected, (Gp 1 n:1, Gp 2 n:1) and 1 patient declined 1 aspiration (Gp 3 n:1) preventing analysis on these patients.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 9 | 9 | 10 | 12
pg/mL | -1.08 (2.87) | 0.75 (1.98) | -0.28 (0.37) | -0.19 (0.29)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = 0.13, Kruskal-Wallis

5. Secondary Outcome: Synovial Interleukin-1 Receptor Antagonist (IL-1ra) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure IL-1ra concentration using an immunoassay. Data will be presented as the change in IL-1ra concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: Two other patients had dry knee aspirations, where the aspiration was performed but no fluid was collected, (Gp 1 n:1, Gp 2 n:1) and 1 patient declined the pre-op assessment aspiration (Gp 3 n:1) preventing analysis on these patients.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12
pg/mL | -3352.5 (8285.5) | -4955.6 (12,939.6) | -7278.4 (12,581.9) | -6888.5 (8364.2)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = 0.15, Kruskal-Wallis

6. Secondary Outcome: Synovial C-terminal Peptide II (CTXII) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure CTXII concentration using an immunoassay. Data will be presented as the change in CTXII concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: Two other patients had dry knee aspirations, where the aspiration was performed but no fluid was collected, (Group 1 n:1, Group 2 n:1) and 1 patient declined the pre-op assessment aspiration (Group 3 n:1) preventing analysis on these patients.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12
ng/mL | 0.32 (0.21) | 0.23 (0.27) | 0.19 (0.34) | 1.32 (1.10)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = .003, Kruskal-Wallis

7. Secondary Outcome: Synovial Cartilage Oligomeric Matrix Protein (COMP) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure COMP concentration using an immunoassay. Data will be presented as the change in COMP concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12
μg/mL | -4.9 (17.5) | -21.7 (24.1) | -11.7 (7.1) | -22.1 (5.7)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = .007, Kruskal-Wallis

8. Secondary Outcome: Synovial Glycosaminoglycans (GAG) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure GAG concentration using an immunoassay. Data will be presented as the change in GAG concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12
μg/mL | -73.1 (176.7) | 155.8 (132.4) | -49.0 (252.5) | -167.4 (140.0)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = .63, Kruskal-Wallis

9. Secondary Outcome: Synovial Type I Collagen Cross-Linked N-Telopeptide (NTX-I) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure NTX-I concentration using an immunoassay. Data will be presented as the change in NTX-I concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12
µg/mL | 3.5 (7.7) | 0.6 (4.0) | 2.6 (3.6) | 5.8 (6.5)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = 0.17, Kruskal-Wallis

10. Secondary Outcome: Synovial TNF-stimulated Gene 6 Protein (TSG-6) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure TSG-6 concentration using an immunoassay. Data will be presented as the change in TSG-6 concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12
ng/ml | 68.0 (266.0) | 57.6 (244.5) | 111.4 (180.5) | -4.9 (224.0)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = .62, Kruskal-Wallis

11. Secondary Outcome: Synovial Matrix Metalloproteinase 1 (MMP-1) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure MMP-1 concentration using an immunoassay. Data will be presented as the change in MMP-1 concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12
ng/mL | 249.0 (745.9) | -183.0 (245.5) | -395.5 (472.2) | -100.4 (557.9)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = .02, Kruskal-Wallis

12. Secondary Outcome: Synovial Matrix Metalloproteinase 3 (MMP-3) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure MMP-3 concentration using an immunoassay. Data will be presented as the change in MMP-3 concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12
ng/mL | 2702.9 (3937.2) | 504.0 (1705.9) | -512.4 (2175.0) | 1295.9 (2414.3)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = .20, Kruskal-Wallis

13. Secondary Outcome: Synovial Matrix Metalloproteinase 9 (MMP-9) Concentration
Description: Participants will have a knee joint aspiration during their initial orthopedic consult and during pre-op assessment. Synovial fluid will be aspirated and spun at 3500RPM for 10 minutes then the supernatant will be pipetted and frozen. The supernatant will be used to measure MMP-9 concentration using an immunoassay. Data will be presented as the change in MMP-9 concentration from knee aspirate collected during the initial orthopedic consult after injury and during the participant's pre-operative assessment, usually 1-7 days after the initial consult.
Time Frame: Up to seven days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 12
ng/mL | -71.1 (15.9) | -28.9 (42.6) | -17.7 (18.8) | -14.0 (24.5)
Statistical Analysis 1: Comparison: Kenalog or Placebo vs Kenalog Then Placebo vs Kenalog Only vs Placebo; Test type: Superiority; p = .87, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Over the course of 12months.
Description: Patients were approached and asked about any adverse events at regular study and/or clinic visits.
Arm/Group | Kenalog or Placebo | Kenalog Then Placebo | Kenalog Only | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 7/11 | 4/11 | 6/11 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kenalog or Placebo (N=11) | Kenalog Then Placebo (N=11) | Kenalog Only (N=11) | Placebo (N=12)
Nausea or Hives/Rash from post op pain meds (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ACL Re-Tear (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) — Re-Tear of the anterior cruciate ligament
Knee Effusion Post-Op (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Knee Effusion from Unanticipated Accident (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arthrofibrosis (General disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Cervical Strain after Motor Vehicle Accident (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nosebleed (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infrapatella scarring/pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Strep Throat (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Persistent Low Leg Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stitch Abscess (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT01692756/Prot_SAP_000.pdf